CLINICAL TRIAL: NCT01872572
Title: A Phase 1 Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RB006 Administered Subcutaneously, With and Without IV RB007, in Healthy Young Volunteers
Brief Title: Safety, Tolerability and PK/PD of RB006 in a Healthy Volunteer SAD
Acronym: SC101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: REG1-CLINSC101
Record Dates: First submitted 2013-06-02; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Other): Cohort 1: 6 subjects received Subcutaneous RB006 0.5 mg/kg and 2 subjects received SC placebo
  Interventions: Drug: Subcutaneous RB006 0.5 mg/kg; Drug: Placebo
- Cohort 1-A (Other): Cohort 1-A: 4 subjects received open-label Subcutaneous RB006 0.5 mg/kg
  Interventions: Drug: Subcutaneous RB006 0.5 mg/kg
- Cohort 2 (Other): Cohort 2: 6 subjects received Subcutaneous RB006 1.0 mg/kg and 2 subjects received SC placebo
  Interventions: Drug: Subcutaneous RB006 1.0 mg/kg; Drug: Placebo
- Cohort 3 (Other): Cohort 3: 6 subjects received Subcutaneous RB006 3.0 mg/kg and 2 subjects received SC placebo
  Interventions: Drug: Subcutaneous RB006 3.0 mg/kg; Drug: Placebo
- Cohort 4 (Other): 8 subjects received subcutaneous RB006 2.0 mg/kg as well as the following:
  * 4 subjects received an IV bolus injection of 1 mg/kg RB007 at 72 hours post-RB006 administration
  * 4 subjects received an IV bolus injection of 1 mg/kg RB007 at 24, 72, and 120 hours post-RB006 administration
  Interventions: Drug: Subcutaneous RB006 2.0 mg

INTERVENTIONS:
Drug: Subcutaneous RB006 0.5 mg/kg — Subcutaneous RB006 0.5 mg/kg
  Other Names: SC RB006
  Arms: Cohort 1; Cohort 1-A
Drug: Subcutaneous RB006 1.0 mg/kg — Subcutaneous RB006 1.0 mg/kg
  Other Names: SC RB006
  Arms: Cohort 2
Drug: Subcutaneous RB006 3.0 mg/kg — Subcutaneous RB006 3.0 mg/kg
  Other Names: SC RB006
  Arms: Cohort 3
Drug: Subcutaneous RB006 2.0 mg — * Arm 1: 4 subjects received an IV bolus injection of 1 mg/kg RB007 at 72 hours post-RB006 administration
  * Arm 2: 4 subjects received an IV bolus injection of 1 mg/kg RB007 at 24, 72, and 120 hours post-RB006 administration.
  Other Names: SC RB006
  Arms: Cohort 4
Drug: Placebo — Placebo
  Other Names: SC Placebo
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
This was a Phase 1a, single-center, double-blind, randomized, placebo-controlled study of the safety, tolerability, PK, and PD of single ascending doses of RB006 administered as an SC injection, with and without IV RB007 (an active control agent for RB006), in healthy young volunteers. The study originally planned to enroll 4 cohorts of 8 subjects each (N=32); however, upon review cohort (Cohort 1-A) was necessary in order to fully define the PK profile of SC RB006. Therefore, 36 subjects were enrolled in this study.

Each cohort was balanced by sex with no more than 2/3 of one sex enrolled in any particular cohort (i.e., 5 of 8 subjects in each cohort). No subject participated in >1 dose group, and progression to the next higher dose only occurred if the prior dose level was well tolerated, as assessed by a Safety Review Committee (SRC)

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB)-approved informed consent was signed and dated prior to any study-related activities.
2. Subject was between the ages of 18 and 45 years, inclusive.
3. Subject was a female with a negative urine or serum pregnancy test or postmenopausal for at least 1 year prior to randomization.
4. Subject had a body mass index (BMI) between 18 kg/m2 and 32 kg/m2 (weight/[height]2) and was ≥50 kg and ≤120 kg total body weight.
5. Subject had normal (or abnormal and clinically insignificant) laboratory values at Screening.
6. Subject was medically normal with no significant abnormal findings at the Screening physical examination.
7. Subject had the ability to understand the requirements of the study and a willingness to comply with all study procedures.
8. Subject had not consumed and agreed to abstain from taking any dietary supplements or nonprescription drugs
9. Subject had not consumed and agreed to abstain from taking any prescription drugs
10. Subject had not consumed alcohol-containing beverages for 3 days prior to CRU admission
11. Subject had not consumed grapefruit or grapefruit juice within the 14 days prior to CRU admission
12. Subject had not used tobacco or nicotine-containing products within 6 months prior to CRU admission

Exclusion Criteria:

1. Evidence or history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal (GI), cardiovascular, hematologic, metabolic, neurological, immunologic, nephrologic, endocrine, or psychiatric disease.
2. Any evidence or history of intracranial bleeding, aneurysm, or thrombotic or hemorrhagic stroke.
3. Any known individual or family history of a bleeding diathesis or coagulopathy.
4. Active or expected menstruation during the Treatment Phase (females only).
5. History of thrombocytopenia associated with abnormal bleeding or risk of a bleeding event, or screening or baseline platelet count <100,000/mm3.
6. History of thrombocytosis associated with a thrombotic event or risk for a thrombotic event, or screening or baseline platelet count >600,000/mm3.
7. Endoscopically confirmed peptic ulcer disease within 3 years of CRU admission or GI bleeding within 3 months of CRU admission, including a positive stool for occult blood at Screening or Baseline.
8. Urinary tract bleeding within 3 months of CRU admission, including microscopic hematuria on screening or baseline urinalysis.
9. Unusual or prolonged bleeding (e.g., gum bleeding, nosebleeds, easy bruising), as documented on the Self-Reported Bleeding Questionnaire, at Screening.
10. Severe trauma, fracture, major surgery, or biopsy of a parenchymal organ within 3 months of CRU admission.
11. Severe persistent hypertension (systolic pressure >180 mmHg or diastolic pressure >110 mmHg).
12. Baseline hemoglobin <12.0 g/dL for males or <11.0 g/dL for females; prothrombin time (PT) greater than the ULN; or aPTT greater than the ULN.
13. Clinically significant liver dysfunction (e.g., as evidenced by elevated liver function tests).
14. Clinically significant renal dysfunction (e.g., estimated glomerular filtration rate <60 mL/min or serum creatinine >1.5 mg/dL).
15. History of illicit drug abuse in the past year or current evidence of such abuse in the opinion of the Investigator.
16. Positive findings on urine drug screen.
17. Positive findings for human immunodeficiency virus, hepatitis B, and/or hepatitis C at Screening.
18. Pregnant or lactating.
19. Acute illness within 1 week of CRU admission.
20. A history of alcohol abuse in the past year relative to CRU admission.
21. Donated plasma within 7 days of study drug administration.
22. Donated 1 or more pints of blood (or equivalent blood loss) within 6 weeks prior to study drug administration.
23. Use of an investigational drug within 30 days prior to CRU admission or prior REG1 Anticoagulation System exposure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Primary Outcome of this study using SC RB006 with and without RB007 in healthy volunteers was safety as determined by Treatment Emergent Adverse Events | 10 days

SECONDARY OUTCOMES:
Outcome of this study using SC RB006 with and without RB007 in healthy volunteers was safety as determined by Serious Adverse Events | 10 days
Outcome of this study using SC RB006 with and without RB007 in healthy volunteers was pharmacodynamics as determined by change from baseline in aPTT | Pre-dose, 1, 2, 3, 6, 9, 12, 15, 18, 24, 30, 36, 48, 60, 72, 84, 96, 120, 144, 168, 216 (and if applicable, 264) hours post RB006 dose
Outcome of this study using SC RB006 with and without RB007 in healthy volunteers was pharmacokinetics as determined by Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 1, 2, 3, 6, 9, 12, 15, 18, 24, 30, 36, 48, 60, 72, 84, 96, 120, 144, 168, and 216 (and if applicable, 264) hours post-RB006 dose

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Medlock, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- [Result] Vavalle JP, Rusconi CP, Zelenkofske S, Wargin WA, Alexander JH, Becker RC. A phase 1 ascending dose study of a subcutaneously administered factor IXa inhibitor and its active control agent. J Thromb Haemost. 2012 Jul;10(7):1303-11. doi: 10.1111/j.1538-7836.2012.04742.x. PMID 22500821
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581